CLINICAL TRIAL: NCT03961256
Title: A Phase 2, Prospective, Randomized, Multicenter, Open-Label, Controlled Trial to Assess the Efficacy and Safety of Exenatide SR for the Prevention of Diabetes After Kidney Transplantation.
Brief Title: Assess the Efficacy and Safety of Exenatide SR for the Prevention of Diabetes After Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Stegall, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-000649
Record Dates: First submitted 2019-04-23; First posted 2019-05-23 (Actual); Results first posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Pre Diabetes
Keywords: Kidney Transplant
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exenatide SR Intervention Group (Experimental): Subjects will receive, in addition to standard care, Exenatide SR 2 mg subcutaneous (SQ) weekly for 24 months.
  Interventions: Drug: Exenatide SR
- Standard of Care (No Intervention): Subjects will receive standard post-transplant care as per Mayo Clinic usual practice.

INTERVENTIONS:
Drug: Exenatide SR — Exenatide SR 2 mg subcutaneous (SQ) weekly
  Arms: Exenatide SR Intervention Group

SUMMARY:
Researchers are trying to determine if an anti-diabetes medication, called Exenatide SR, is well tolerated in kidney transplant patients with elevated blood glucose levels, and if it's effective in preventing diabetes.

DETAILED DESCRIPTION:
New diabetes can develop after transplant and may affect a transplanted kidney's health and a recipient's overall health. Currently, patients who are pre-diabetic are encouraged to exercise and lose weight. Researchers are planning to test whether an addition of this medication will lead to better results and more effectively prevent diabetes in patients who already have high blood sugars.

Exenatide SR is medication given by weekly injection. It increases insulin release in response to a meal and slows digestion. This medicine is already in use and approved by the US Food and Drug Administration (FDA) in patients with diabetes. However, it has not been approved for this indication; the FDA has allowed the use of this drug in this research study.

ELIGIBILITY:
Inclusion criteria:

* Recipients of solitary kidney transplants (i.e. not combined liver-kidney, pancreas-kidney etc.)
* At 4 months after transplantation: Prediabetes (fasting blood glucose 100-125 mg/dl; or 2 hr glucose 140-199 or HgbA1c 5.7-6.4%)

Exclusion criteria:

* Diabetes pre-transplantation
* Diabetes at 4 months
* <18 years of age
* eGFR <30 ml/min (estimated by MDRD equation from serum creatinine)
* Active acute cellular rejection including borderline (If treated and resolved, these patients can be included)
* BK nephropathy active
* History of pancreatitis, pre-existing moderate-to-severe gastroparesis, liver cirrhosis or family /personal history of multiple endocrine neoplasia 2 or medullary thyroid cancer
* Pregnant or breastfeeding women. Female Subject must be either:

  * Of non-child bearing potential: Post-menopausal (defined as at least 1 year without any menses) prior to screening , or documented surgically sterile or status post-hysterectomy
  * Or if childbearing potential, agree not to try and become pregnant during the study for at least 90 days after the final study drug administration. And have a negative serum or urine pregnancy test. And if heterosexually active, agree to consistently use two forms of highly effective birth control.
* Hypersensitivity to Exenatide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Stegall, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide SR Intervention Group: Subjects received, in addition to standard care, Exenatide SR 2 mg subcutaneous (SQ) weekly for 24 months.
  Exenatide SR: Exenatide SR 2 mg subcutaneous (SQ) weekly
- Standard of Care: Subjects received standard post-transplant care as per Mayo Clinic usual practice.
Period: Overall Study
Arm/Group | Exenatide SR Intervention Group | Standard of Care
Started | 6 | 3
Completed | 6 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide SR Intervention Group | Standard of Care | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48.5 [39.0 to 54.1] | 57.7 [42.5 to 59.2] | 53.5 [37.5 to 57.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression From Prediabetes to Diabetes
Description: Number of subjects to have an increase in HbA1C or fasting blood sugar to diabetic range based on the American Diabetes Association (ADA) criteria after kidney transplantation
Time Frame: 12 months after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide SR Intervention Group | Standard of Care
Number analyzed (Participants) | 6 | 3
Participants | 0 | 1

2. Secondary Outcome: Progression From Prediabetes to Diabetes
Description: as for outcome 1
Time Frame: 24 months after transplantation
Population: Data was not collected nor analyzed for one subject in the standard of care arm
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide SR Intervention Group | Standard of Care
Number analyzed (Participants) | 6 | 2
Participants | 1 | 1

3. Secondary Outcome: Creatinine
Description: A creatinine blood test measures the level of creatinine in the blood. Creatinine is a waste product that forms when creatine, which is found in the muscle, breaks down. Creatinine levels in the blood can provide the doctors with information about how well the kidneys are working. As measured in mg/dL units.
Time Frame: From enrollment, up to 20 months post-enrollment
Population: Data was not collected nor analyzed for one subject in the standard of care arm
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Exenatide SR Intervention Group | Standard of Care
Number analyzed (Participants) | 6 | 2
mg/dL | 1.7 [1.5 to 1.9] | 1.4 [1.2 to 1.6]

4. Secondary Outcome: Hemoglobin A1c
Description: Hemoglobin is a protein within red blood cells. As glucose enters the bloodstream, it binds to hemoglobin, or glycates. The more glucose that enters the bloodstream, the higher the amount of glycated hemoglobin. An A1C level below 5.7 percent is considered normal.
Time Frame: 12 and 24 months after kidney transplantation
Population: Data was not collected nor analyzed for one subject in the standard of care arm
Measure: Median (Inter-Quartile Range); unit: percentage of glycated hemoglobin
Arm/Group | Exenatide SR Intervention Group | Standard of Care
Number analyzed (Participants) | 6 | 2
percentage of glycated hemoglobin
  12 months | 5.6 [5.3 to 5.8] | 5.85 [5.3 to 6.4]
  24 months | 5.65 [5.6 to 6.7] | 5.75 [5.3 to 6.2]

5. Secondary Outcome: Incidence of Mesangial Expansion
Description: Number of subjects to experience mesangial expansion >20%. Mesangial expansion occurs due to increased deposition of extracellular matrix proteins, for example fibronectin, into the mesangium. Accumulation of extracellular matrix proteins then occurs due to insufficient degradation by matrix metalloproteinases.
Time Frame: 12 and 24 months after kidney transplantation
Population: Data was not collected nor analyzed for one subject in the standard of care arm at 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide SR Intervention Group | Standard of Care
Number analyzed (Participants) | 6 | 3
Participants
  12 months | 0 | 0
  24 months: number analyzed (Participants) | 6 | 2
  24 months | 0 | 0

6. Secondary Outcome: Incidence of Death
Description: Number of subjects to experience death by any cause
Time Frame: From enrollment, up to 20 months post-enrollment
Population: Deaths collected for the Exenatide SR Intervention Group only. Deaths were not collected for the Standard of Care arm
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide SR Intervention Group
Number analyzed (Participants) | 6
Participants | 0

7. Secondary Outcome: Graft Loss
Description: The number of subjects to experience graft loss. Primary graft failure is defined as no evidence of engraftment or hematological recovery of donor cells, within the first month after transplant, without evidence of disease relapse. Secondary graft failure refers to the loss of a previously functioning graft, resulting in cytopenia involving at least two blood cell lineages.
Time Frame: From enrollment, up to 20 months post-enrollment
Population: Graft loss collected for the Exenatide SR Intervention Group only. Graft Loss was not collected for the Standard of Care arm
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide SR Intervention Group
Number analyzed (Participants) | 6
Participants | 0

8. Secondary Outcome: Adverse Events for Exenatide SR Intervention
Description: Total number of adverse events reported by the subjects that received the Exenatide SR Intervention
Time Frame: 12 months
Measure: Number; unit: Adverse Events
Arm/Group | Exenatide SR Intervention Group
Number analyzed (Participants) | 6
Adverse Events | 10

ADVERSE EVENTS:
Time Frame: Deaths were assessed up to 20 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were assessed up to 12 months.
Description: Deaths and Adverse Events collected for the Exenatide SR Intervention Group only. Deaths and Adverse Events were not collected for the Standard of Care arm
Arm/Group | Exenatide SR Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide SR Intervention Group (N=6)
Nausea (General disorders) | 1
Vomiting (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Abdominal pain (General disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT03961256/Prot_SAP_000.pdf